CLINICAL TRIAL: NCT05023356
Title: Non-contact Vital Signs Monitoring in Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-05-024CC
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; Vital Signs; Monitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contact vital signs monitoring: Routine monitors with cables
- Non-contact vital signs monitoring: Camera
  Interventions: Device: Non-contact vital signs monitoring with camera

INTERVENTIONS:
Device: Non-contact vital signs monitoring with camera — Monitor patients face image by non-contact vital signs monitoring with camera
  Groups: Non-contact vital signs monitoring

SUMMARY:
The purpose of this study is to monitor vital signs with contact and non-contact monitors in patients during anesthesia, and analyze the signal differences between the two monitors.

DETAILED DESCRIPTION:
The standard vital signs routinely monitored in patients during anesthesia include heart rate, electrocardiogram, blood pressure, body temperature, respiratory rate, and peripheral blood oxygen saturation, and etc. Continuous measurement and interpretation of these vital signs can provide important information about the underlying physiological state.

Conventional techniques for tracking vital signs require physical contact, and most techniques are invasive. Body contact with sensors (for example, electrocardiograph electrodes) can irritate or damage the patient's skin, interfere with the patient's treatment or comfort, provide a vector for infection and cross-contamination, and only hinder mobility. In addition, when placing the sensor/wire on the body, the patient may feel uncomfortable (for example, anxiety, tension, and excitement). This negative experience may change the patient's breathing and heart rate and produce misleading results for medical service providers. Therefore, people need effective sensing methods that can wirelessly (non-contact/remote) monitor vital signs.

Since the 1970s, researchers have been looking for ways to conduct non-contact monitoring of vital signs. The following important medical situations have promoted continuous research in this field: (1) The patient's skin is fragile or vulnerable, such as low birth weight. , Premature infants, burn patients; (2) monitor wiring can endanger or interfere with patients, such as: Infant Death Syndrome and sleep apnea; (3) cross-contamination between patients (such as reusable wires) . The non-contact life monitoring technology does not involve electrodes or adhesives, does not touch the skin, does not have the risk of wires, entanglements or patient discomfort, does not consume any consumables, and there is no chance of cross-infection caused by inadequately disinfected equipment.

Today, advances in sensing technology have enabled smart systems to monitor vital signs, such as respiration and heart rate, in a non-contact manner. The two most advanced non-contact vital signs monitoring methods are the use of radio frequency (radar) and imaging (camera). In the past 15 years, the development of camera technology has increased its applicability and affordability, making people more and more interested in using these technologies in medical institutions. Monitoring methods using images can measure multiple vital signs at the same time and are relevant. The research has been applied to many ethnic groups, including sleeping healthy people, intensive care unit patients, kidney dialysis patients, and fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 20.
* American Society of Anesthesiologists (American Society of Anesthesiologists, ASA) anesthesia risk class l (healthy people, except for the surgical correction part, no systemic disease, mortality before and after surgery 0.06~0.08%) and ASA class II patients (with mild systemic disease but no functional impairment, and the mortality rate before and after surgery is 0.27~0.4%).

Exclusion Criteria:

* under the age of 20
* pregnant patients
* those who refuse to participate in the research or are unwilling to sign the consent form due to any factors

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 20, ASA class I~II who accept scheduled anesthesia and surgery in single medical center are enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-10 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-05-23 (Estimated)

PRIMARY OUTCOMES:
Signal similarities | During anesthesia procedure
  After analyzing signals from contact and non-contact vital signs monitors in the same group of patients in anesthesia, we could find out some signal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chuan Kuo, PhD, Principal Investigator — Institute of Biophotonics, National Yang Ming Chiao Tung University, Taiwan; Chien-Kun Ting, PhD, Principal Investigator — Department of Anesthesiology, Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be constructed for business model.

REFERENCES:
- [Background] Matthews G, Sudduth B, Burrow M. A non-contact vital signs monitor. Crit Rev Biomed Eng. 2000;28(1-2):173-8. doi: 10.1615/critrevbiomedeng.v28.i12.290. PMID 10999382
- [Background] Luo J, Yan Z, Guo S, Chen W. Recent Advances in Atherosclerotic Disease Screening Using Pervasive Healthcare. IEEE Rev Biomed Eng. 2022;15:293-308. doi: 10.1109/RBME.2021.3081180. Epub 2022 Jan 20. PMID 34003754
- [Background] Chen KM, Misra D, Wang H, Chuang HR, Postow E. An X-band microwave life-detection system. IEEE Trans Biomed Eng. 1986 Jul;33(7):697-701. doi: 10.1109/TBME.1986.325760. No abstract available. PMID 3733127